CLINICAL TRIAL: NCT04021238
Title: Contrast-Enhanced Ultrasound for Kidney Cancer Subtyping and Staging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC1922
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Perflutren Lipid Microsphere or Lumason (Experimental): Patients with suspected kidney cancer and planned surgery will be imaged using contrast-enhanced ultrasound with either perflutren or Lumason.
  Interventions: Drug: Perflutren lipid microsphere; Drug: Sulfur hexafluoride lipid microspheres

INTERVENTIONS:
Drug: Perflutren lipid microsphere — Baseline B-mode US will be performed to confirm the lesions being imaged (unless it is a subject with no lesions, then a basic B-mode US will be performed. Perflutren is a diagnostic drug that is intended to be used for contrast enhancement. The vial contains a clear, colorless, sterile, non-pyrogenic, hypertonic solution which is activated by mechanical agitation with Vialmix®.It will be dispensed in inactivated form to a study team member. The contrast agent will be activated just prior to administration (ideally to be used within 5 minutes of activation). Contrast agent Definity (or Lumason) will be activated according to package insert instructions, including use of VialMix®, the device used to activate Definity. Administration will occur IV in coordination with sonography staff trained specifically in contrast ultrasound imaging.The total imaging time is anticipated to be less than 30 minutes.
  Other Names: Definity; Microbubble contrast agent
Drug: Sulfur hexafluoride lipid microspheres — Baseline B-mode US will be performed to confirm the lesions being imaged (unless it is a subject with no lesions, then a basic B-mode US will be performed. Lumason will be used as a secondary contrast agent only if Definity(perflutren) is unavailable.This drug will be administered using the dosing range and administration type within the Lumason prescribing information. The contrast agent will be activated just prior to administration (ideally to be used within 5 minutes of activation). Contrast agent Definity (or Lumason) will be activated according to package insert instructions, including use of VialMix®, the device used to activate Definity. Administration will occur IV in coordination with sonography staff trained specifically in contrast ultrasound imaging.The total imaging time is anticipated to be less than 30 minutes.
  Other Names: Lumason

SUMMARY:
The purpose of this study is to determine if contrast-enhanced ultrasound can detect abnormal features of kidney lesions in patients with suspected kidney cancer with the same accuracy as conventional ultrasound and contrast-enhanced magnetic resonance imaging (MRI)

DETAILED DESCRIPTION:
This is a pilot cross-sectional study that compares contrast enhanced ultrasound to conventional ultrasound and contrasted MRI. Eligible patients will include anyone who has suspected kidney cancer and is scheduled for surgery, up to an anticipated total of 40 participants. Subject participation will be only for the day of CEUS study. There will be no follow-up period for this study. However, if results are encouraging, a longitudinal observational study may follow, and these same subjects would be eligible for enrollment. Eligible subjects will undergo a contrast enhanced ultrasound.

Following completion of imaging, all CEUS, MRI (within 4 months) and B-mode (at time of CEUS) US studies will be de-identified. Blinded radiologists will interpret images and provide an overall assessment of risk of malignancy to each kidney using the Bosniak criteria for each kidney lesion present. The Bosniak criteria places cystic lesions into one of 5 categories (I, II, IIF, III and IV) based on lesion characteristics. CEUS based diagnosis will be compared to the diagnoses on routine B-mode US and contrast-enhanced MRI.

ELIGIBILITY:
Inclusion Criteria:

* A suspected diagnosis of kidney cancer with a solid or partially solid lesion and planned surgical nephrectomy within 3 months before surgery
* Able to provide informed consent
* Willing to comply with protocol requirements
* At least 18 years of age

Exclusion Criteria:

* Critically ill or medically unstable or in an intensive care setting and whose critical course during a potential observation period would be unpredictable
* Known hypersensitivity to sulfur hexafluoride or to any component of perflutren lipid (Definity®) or sulfur hexafluoride (Lumason®)
* Right to left shunt, severe pulmonary hypertension (Pulmonary artery pressure >90mmHg), or adult respiratory distress syndrome
* Has any other medical condition or other circumstances that would significantly decrease the chances of obtaining reliable data or of achieving the study objectives
* Unstable cardiopulmonary disease including any of the following:

  * Severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association)
  * Unstable angina
  * Symptomatic arrhythmia (i.e. tachycardia, bradycardia, supraventricular tachycardia, ventricular fibrillation, ventricular tachycardia, atrial flutter or fibrillation)
  * Myocardial infarction within 14 days prior to the date of proposed microbubble administration.
* Any woman who is pregnant or has reason to believe she is pregnant (the possibility of pregnancy has to be excluded by negative urine β-HCG results, obtained the same day as the CEUS, or on the basis of patient history, e.g.: tubal ligation, hysterectomy or a minimum of 1 year without menses)
* Obesity that limits obtainment of acceptable images

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chang, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 10/7/2020- 7/22/2022, 25 subjects consented and enrolled in the study at one center in North Carolina.
Pre-assignment Details: A total of 25 subjects were found eligible and consented to the study. One subject was withdrawn after enrollment and did not complete study imaging and 24 subjects enrolled in the study and underwent research imaging.
Groups:
- Perflutren Lipid Microsphere: Subjects with suspected kidney cancer and planned surgery were imaged using Definity® containing perflutren lipid microsphere contrast-enhanced ultrasound (US). Baseline B-mode US was performed to confirm the lesions being imaged.
Period: Overall Study
Arm/Group | Perflutren Lipid Microsphere
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects with suspected kidney cancer and planned surgery.
Groups:
- Perflutren Lipid Microsphere or Lumason: Subjects with suspected kidney cancer and planned surgery were imaged using Definity® containing perflutren lipid microsphere contrast-enhanced ultrasound (US). Baseline B-mode US was performed to confirm the lesions being imaged.
Arm/Group | Perflutren Lipid Microsphere or Lumason
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: 3D CEUS Generated Metrics in Kidney Mass: Wash_In_Slope
Description: A study-specific model was created to predict kidney tumor type. The contrast-enhanced ultrasonogram (CEUS) Wash_In_Slope parameter was generated. This metric indicates the change in contrast with time in the mass using bolus imaging. Bolus imaging injects a small amount of contrast agent and monitors the contrast agent as it flows in (wash-in) and out (wash-out) of the body/mass. The intensity of the signal (the brightness of the image) is plotted over time to generate the time-intensity curve. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White.The Wash_In_Slope increases as the contrast agent is introduced to the body/mass. This value was generated by fitting the data to a linear equation. Increasing brightness is related to the slope of curve.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: AU/second
Groups:
- CEUS Imaging Parameters: CEUS-generated parameters : Wash_In_Slope generated from MATLAB for the analysis.
Arm/Group | CEUS Imaging Parameters
Number analyzed (Participants) | 14
AU/second | 7.60 [3.13 to 12.28]

2. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass: Wash_In_intercept
Description: A study-specific model was created to predict kidney tumor type. The contrast-enhanced ultrasonogram (CEUS) Wash_In_intercept parameter was generated. This metric indicates the intensity level prior to infusion of contrast. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=white. This value was calculated using an equation for a line which has a slope and the intercept. The values were negative because they were calculated (not measured).
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: Units on a scale
Groups:
- CEUS Imaging Parameters: CEUS-generated parameters : Wash_In_intercept generated from MATLAB for the analysis.
Arm/Group | CEUS Imaging Parameters
Number analyzed (Participants) | 14
Units on a scale | -18.30 [-149.6 to 62.11]

3. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass: Wash_Out_Slope
Description: A study-specific model was created to predict kidney tumor type. The contrast-enhanced ultrasonogram (CEUS) Wash_Out_Slope parameter was generated. This metric indicates the change in contrast with time in the mass using bolus imaging. Bolus imaging injects a small amount of contrast agent and monitors the contrast agent as it flows in (wash-in) and out (wash-out) of the body/mass. The intensity of the signal (the brightness of the image) is plotted over time to generate the time-intensity curve. The intensity of the signal (the brightness of the image) value range was between 0=black and 255=White. The wash Out slope decreases as the contrast agent clears the body/mass. Decreasing brightness is related to the slope of the curve. This results in a negative number. This value was generated by fitting the data to a linear equation.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: AU/second
Groups:
- CEUS Imaging Parameters: CEUS-generated parameters : , Wash_Out_Slope generated from MATLAB for the analysis.
Arm/Group | CEUS Imaging Parameters
Number analyzed (Participants) | 14
AU/second | -0.93 [-2.09 to -0.41]

4. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass: Wash_Out_Intercept
Description: A study-specific model was created to predict kidney tumor type. The contrast-enhanced ultrasonogram (CEUS) Wash_Out_Intercept parameter was generated. This metric indicates the intensity level of contrast at a steady state of enhancement in the mass. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White. This value was calculated using an equation for a line that has a slope and an intercept.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- CEUS Imaging Parameters: CEUS-generated parameters : Wash_Out_Intercept generated from MATLAB for the analysis.
Arm/Group | CEUS Imaging Parameters
Number analyzed (Participants) | 14
units on a scale | 125.84 [43.28 to 199.71]

5. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass: FR_a
Description: A study-specific model was created to predict kidney tumor type. The contrast-enhanced ultrasonogram (CEUS) FR_a parameter was generated. The intensity of the signal (the brightness of the image) value range is between 0=black, and 255=white. The intensity was plotted by time. FR_a parameters were devised from an exponential fit. The exponential fit of the data provides the height of the curve.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: Units on a scale
Groups:
- CEUS Imaging Parameters: CEUS-generated parameters : FR_a generated from MATLAB for the analysis.
Arm/Group | CEUS Imaging Parameters
Number analyzed (Participants) | 14
Units on a scale | 102.84 [61.01 to 152.8]

6. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass: FR_beta
Description: A study-specific model was created to predict kidney tumor type. The contrast-enhanced ultrasonogram (CEUS) FR_beta parameter was generated. The intensity of the signal (the brightness of the image) value range is between 0=black, 255=White. The intensity was plotted by time. FR_beta parameters were devised from an exponential fit. Exponential fit of the data provides the slope of the curve.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: AU/second
Groups:
- CEUS Imaging Parameters: CEUS-generated parameters : FR_beta generated from MATLAB for the analysis.
Arm/Group | CEUS Imaging Parameters
Number analyzed (Participants) | 14
AU/second | 0.16 [0.03 to 0.77]

7. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass: Volume
Description: A study-specific model was created to predict kidney tumor type. The contrast-enhanced ultrasonogram (CEUS) volume parameter was generated. The volumes were generated using the ellipsoid equation on the CEUS image of the kidney mass.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: milliliters
Groups:
- CEUS Imaging Parameters: CEUS-generated parameters: Volume generated from MATLAB for the analysis.
Arm/Group | CEUS Imaging Parameters
Number analyzed (Participants) | 14
milliliters | 60.80 [3.08 to 271.97]

8. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass - Histopathologic Type vs. Wash_In_Slope
Description: The association between tumor pathology type (Clear cell renal carcinoma (CCRCC) versus none (CCRCC) pathology) and CEUS-generated Wash_In_Slope parameter was studied. This metric indicates the change in contrast intensity with time in the mass using bolus imaging. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White. The Wash_In_Slope increases as the contrast agent is introduced to the body/mass. This value was generated by fitting the data to a linear equation. Increasing brightness is related to the slope of the curve.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Deviation); unit: AU/second
Groups:
- Clear Cell Renal Carcinoma: Clear cell renal carcinoma type
- Papillary Carcinoma: papillary carcinoma type
- Clear Cell Papillary: Clear cell papillary type
- Chromophobe: chromophobe type
- Other: other type
Arm/Group | Clear Cell Renal Carcinoma | Papillary Carcinoma | Clear Cell Papillary | Chromophobe | Other
Number analyzed (Participants) | 10 | 1 | 1 | 1 | 1
AU/second | 7.61 (2.33) | 3.13 (NA) — Only 1 subject | 4.23 (NA) — Only 1 subject | 10.56 (NA) — Only 1 subject | 12.28 (NA) — Only 1 subject

9. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass - Histopathologic Type vs. Wash_In_intercept
Description: The association between tumor pathology type (Clear cell renal carcinoma (CCRCC) versus none (CCRCC) pathology) and CEUS-generated Wash_In_intercept parameter was studied. This metric indicates the intensity level prior to infusion of contrast. The intensity of the signal (the brightness of the image) value range is between 0=black, and 255=White. This value was calculated using an equation for a line which has a slope and the intercept. The values were negative because they were calculated (not measured).
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Clear Cell Renal Carcinoma | Papillary Carcinoma | Clear Cell Papillary | Chromophobe | Other
Number analyzed (Participants) | 10 | 1 | 1 | 1 | 1
Units on a scale | -11.02 (58.96) | -1.07 (NA) — Only 1 subject | 31.12 (NA) — Only 1 subject | -53.10 (NA) — Only 1 subject | -122.88 (NA) — Only 1 subject

10. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass - Histopathologic Type vs. Wash_Out_Slope
Description: The association between tumor pathology type (Clear cell renal carcinoma (CCRCC) versus none (CCRCC) pathology) and CEUS-generated Wash_Out_Slope parameter was studied. This metric indicates the change in contrast intensity with time in the mass using bolus imaging. The intensity of the signal (the brightness of the image) value range is between 0=black, and 255=White. Decreasing brightness is related to the slope of the curve. The Wash Out slope decreases as the contrast agent clears the body/mass. Decreasing brightness is related to the slope of the curve. This results in a negative number. This value was generated by fitting the data to a linear equation.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Deviation); unit: AU/second
Arm/Group | Clear Cell Renal Carcinoma | Papillary Carcinoma | Clear Cell Papillary | Chromophobe | Other
Number analyzed (Participants) | 10 | 1 | 1 | 1 | 1
AU/second | 7.62 (2.33) | 3.13 (NA) — Only 1 subject | 4.23 (NA) — Only 1 subject | 10.56 (NA) — Only 1 subject | 12.3 (NA) — Only 1 subject

11. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass - Histopathologic Type vs. Wash_Out_Intercept
Description: The association between tumor pathology type (Clear cell renal carcinoma (CCRCC) versus none (CCRCC) pathology) and CEUS-generated Wash_Out_Intercept parameter was studied. This metric indicates the intensity level of contrast at steady state of enhancement in the mass. The contrast-enhanced ultrasonogram (CEUS) Wash_Out_Intercept parameter was generated. The intensity of the signal (the brightness of the image) value range is between 0=black, and 255=White. This value was calculated using an equation for a line which has a slope and the intercept.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Clear Cell Renal Carcinoma | Papillary Carcinoma | Clear Cell Papillary | Chromophobe | Other
Number analyzed (Participants) | 10 | 1 | 1 | 1 | 1
Units on a scale | 137.95 (36.88) | -0.43 (NA) — only 1 subject | 118.53 (NA) — only 1 subject | 139.01 (NA) — only 1 subject | 148.49 (NA) — only 1 subject

12. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass - Histopathologic Type vs. FR_a
Description: The association between tumor pathology type (Clear cell renal carcinoma (CCRCC) versus none (CCRCC) pathology) and CEUS-generated FR_a parameter was studied. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White. The intensity was plotted by time. FR_a parameters were devised from an exponential fit. The exponential fit of the data provides the height of the curve.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Clear Cell Renal Carcinoma | Papillary Carcinoma | Clear Cell Papillary | Chromophobe | Other
Number analyzed (Participants) | 10 | 1 | 1 | 1 | 1
Units on a scale | 105.34 (27.09) | 0 (NA) — only 1 subject | 0 (NA) — only 1 subject | 0 (NA) — only 1 subject | 0 (NA) — only 1 subject

13. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass - Histopathologic Type vs. FR_beta
Description: The association between tumor pathology type (Clear cell renal carcinoma (CCRCC) versus none (CCRCC) pathology) and CEUS-generated FR_ beta parameter was studied. The contrast-enhanced ultrasonogram (CEUS) FR_beta parameter was generated. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White. The intensity was plotted by time. FR_beta parameters were devised from an exponential fit. The exponential fit of the data provides the slope of the curve.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Error); unit: AU/second
Arm/Group | Clear Cell Renal Carcinoma | Papillary Carcinoma | Clear Cell Papillary | Chromophobe | Other
Number analyzed (Participants) | 10 | 1 | 1 | 1 | 1
AU/second | 0.10 (0.06) | 0 (NA) — only 1 subject | 0 (NA) — only 1 subject | 0 (NA) — only 1 subject | 0 (NA) — only 1 subject

14. Primary Outcome: 3D CEUS Generated Metric in Kidney Mass - Histopathologic Type vs. Volume
Description: The association between tumor pathology type (Clear cell renal carcinoma (CCRCC) versus none (CCRCC) pathology) and CEUS-generated volume parameter was studied. The volumes were generated using the ellipsoid equation on the CEUS image of the kidney mass.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Clear Cell Renal Carcinoma | Papillary Carcinoma | Clear Cell Papillary | Chromophobe | Other
Number analyzed (Participants) | 10 | 1 | 1 | 1 | 1
milliliters | 57.93 (81.07) | 260.78 (NA) — only 1 subject | 3.08 (NA) — only 1 subject | 4.77 (NA) — only 1 subject | 3.16 (NA) — only 1 subject

15. Secondary Outcome: 3D CEUS Generated Metric in Kidney Mass - Tumor Stage vs. Wash_In_Slope
Description: The intensity of the signal (the brightness of the image) is plotted over time to generate the time-intensity curve. The intensity of the signal (the brightness of the image) values range between 0=black and 255=White. The Wash_In_Slope increases as the contrast agent is introduced to the body/mass. This value was generated by fitting the data to a linear equation. Increasing brightness is related to the slope of the curve. The association between tumor stage (Tumor stage 0,1,2,3) and CEUS-generated Wash_In_Slope parameter was studied.
  Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to American Joint Cancer Committee. All masses in this study were in stage 0, I, II or III (not stage IV). Stage 0 = cancer cell was not found on pathology. Stage I =tumors size ≤7 cm. Stage II = tumor size >7 cm. Stage III includes tumors that are growing into a major vein or tissue around the kidney with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: AU/second
Groups:
- Stage 0: Disease stage 0
- Stage I; Stage II: Disease stage 2
- Stage III: Disease stage 3
Arm/Group | Stage 0 | Stage I | Stage II | Stage III
Number analyzed (Participants) | 1 | 8 | 3 | 2
AU/second | 12.27 [12.27 to 12.27] | 6.91 [3.51 to 10.57] | 6.72 [3.26 to 9.51] | 9.32 [2.55 to 11.13]

16. Secondary Outcome: 3D CEUS Generated Metric in Kidney Mass - Tumor Stage vs. Wash_In_intercept
Description: The association between tumor stage and CEUS-generated Wash_In_intercept parameter was studied. These values were generated by fitting the data to a linear equation. This metric indicates the intensity level prior to infusion of contrast. The intensity of the signal (the brightness of the image) value range is between 0=black, and 255=White. This value was calculated using an equation for a line that has a slope and an intercept. The values were negative because they were calculated (not measured).
  Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to the American Joint Cancer Committee. All masses in this study were in stage 0, I, II, or III (not stage IV). Stage 0 = cancer cell was not found on pathology. Stage I =tumors size ≤7 cm. Stage II = tumor size >7 cm. Stage III includes tumors that are growing into a major vein or tissue around the kidney with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Stage 0 | Stage I | Stage II | Stage III
Number analyzed (Participants) | 1 | 8 | 3 | 2
Units on a scale | -122.88 [-122.88 to -122.88] | -9.36 [-149.6 to 62] | -25.16 [-69.85 to -1.07] | 8.55 [-1.31 to 18.41]

17. Secondary Outcome: 3D CEUS Generated Metric in Kidney Mass - Tumor Stage vs. Wash_Out_Slope
Description: The association between tumor stage (Tumor stage 0,1,2,3) and CEUS-generated Wash_Out_Slope parameter was studied. The intensity of the signal (the brightness of the image) is plotted over time to generate the time-intensity curve. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White. The Wash_Out_Slope decreases as the contrast agent clears the body/mass. Decreasing brightness is related to the slope of the curve. This results in a negative number. This value was generated by fitting the data to a linear equation. Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to the AJCC. All masses in this study were in stage 0, I, II, or III (not stage IV). Stage 0 = cancer cell was not found on pathology. Stage I =tumors size ≤7 cm. Stage II = tumor size >7 cm, Stage III includes tumors that are growing into a major vein or tissue around the kidney with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: AU/second
Arm/Group | Stage 0 | Stage I | Stage II | Stage III
Number analyzed (Participants) | 1 | 8 | 3 | 2
AU/second | -0.90 [-0.90 to -0.90] | -1.1 [-2.09 to -0.41] | -0.51 [-0.59 to -0.42] | -0.86 [-0.95 to 0.79]

18. Secondary Outcome: 3D CEUS Generated Metric in Kidney Mass - Tumor Stage vs. Wash_Out_Intercept
Description: The association between tumor stage (Tumor stage 0,1,2,3) and CEUS-generated Wash_Out_Intercept parameter was studied. This metric indicates the intensity level of contrast at a steady state of enhancement in the mass. The contrast-enhanced ultrasonogram (CEUS) Wash_Out_Intercept parameter was generated. The intensity of the signal (the brightness of the image) value range is between 0=black, and 255=White. This value was calculated using an equation for a line that has a slope and the intercept.
  Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to the American Joint Cancer Committee. All masses in this study were in stage 0, I, II, or III (not stage IV). Stage 0 = cancer cell was not found on pathology. Stage I =tumors size ≤7 cm. Stage II = tumor size >7 cm. Stage III includes tumors that are growing into a major vein or tissue around the kidney with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Stage 0 | Stage I | Stage II | Stage III
Number analyzed (Participants) | 1 | 8 | 3 | 2
Units on a scale | 148.49 [148.49 to 148.49] | 139.36 [90.17 to 199.71] | 85.72 [43.2 to 122.56] | 154.1 [131.05 to 177.15]

19. Secondary Outcome: 3D CEUS Generated Metric in Kidney Mass - Tumor Stage vs. FR_a
Description: The association between tumor stage (Tumor stage 0,1,2,3) and CEUS-generated FR_a parameter was studied. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White. The intensity was plotted by time. FR_a parameters were devised from an exponential fit. The exponential fit of the data provides the height of the curve.
  Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to the American Joint Cancer Committee. All masses in this study were in stage 0, I, II or III (not stage IV). Stage 0 = cancer cell was not found on pathology. Stage I =tumors size ≤7 cm. Stage II = tumor size >7 cm. Stage III includes tumors that are growing into a major vein or tissue around the kidney with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Stage 0 | Stage I | Stage II | Stage III
Number analyzed (Participants) | 1 | 8 | 3 | 2
Units on a scale | 114.7 [114.7 to 114.7] | 102.8 [61.01 to 152.8] | 86.51 [77.46 to 95.55] | 115.9 [100 to 131.8]

20. Secondary Outcome: 3D CEUS Generated Metric in Kidney Mass - Tumor Stage vs. FR_beta
Description: The association between tumor stage (Tumor stage 0,1,2,3) and CEUS-generated FR_ beta parameter was studied. The contrast-enhanced ultrasonogram (CEUS) FR_beta parameter was generated. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White. The intensity was plotted by time. FR_beta parameters were devised from an exponential fit. The exponential fit of the data provides the slope of the curve.
  Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to the American Joint Cancer Committee. All masses in this study were in stage 0, I, II, or III (not stage IV). Stage 0 = cancer cell was not found on pathology. Stage I =tumors size ≤7 cm. Stage II = tumor size >7 cm. Stage III includes tumors that are growing into a major vein or tissue around the kidney with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: AU/second
Arm/Group | Stage 0 | Stage I | Stage II | Stage III
Number analyzed (Participants) | 1 | 8 | 3 | 2
AU/second | 0.11 [0.11 to 0.11] | 0.20 [0.03 to 0.77] | 0.13 [0.08 to 0.19] | 0.06 [0.03 to 0.09]

21. Secondary Outcome: 3D CEUS Generated Metric in Kidney Mass - Tumor Stage vs. Volume
Description: The association between tumor stage (Tumor stage 0,1,2,3) and CEUS-generated volume was studied. The contrast-enhanced ultrasonogram (CEUS) volume was generated.
  Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to the American Joint Cancer Committee. All masses in this study were in stage 0, I, II or III (not stage IV). Stage 0 = cancer cell was not found on pathology. Stage I =tumors size ≤7 cm. Stage II = tumor size >7 cm. Stage III includes tumors that are growing into a major vein or tissue around the kidney with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Full Range); unit: milliliters
Arm/Group | Stage 0 | Stage I | Stage II | Stage III
Number analyzed (Participants) | 1 | 8 | 3 | 2
milliliters | 3.16 [3.16 to 3.16] | 15.42 [3.07 to 40.7] | 194.43 [50.53 to 271.97] | 70.64 [30.38 to 110.91]

22. Secondary Outcome: Pooled Kidney Mass Stage vs. 3D CEUS-generated Wash in Metrics
Description: The association between pooled tumor stage (tumor stages 0,1,2 versus tumor stage 3) and CEUS-generated Wash_In_Slope parameter was studied. The intensity of the signal (the brightness of the image) is plotted over time to generate the time-intensity curve. The intensity of the signal values range between 0=black and 255=White. The Wash_In_Slope increases as the contrast agent is introduced to the body/mass. This value was generated by fitting the data to a linear equation. Increasing brightness is related to the slope of the curve. Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to the American Joint Cancer Committee. All masses in this study were in stage 0, I, II, or III (not stage IV). Stage 0 = cancer cell was not found on pathology. Stage I =tumors size ≤7 cm. Stage II = tumor size >7 cm. Stage III includes tumors that are growing into a major vein or tissue around the kidney with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Error); unit: AU/second
Groups:
- Stage Non T3: Disease Stage T0, T1 and T2
- Stage T3: Disease Stage T3
Arm/Group | Stage Non T3 | Stage T3
Number analyzed (Participants) | 12 | 2
AU/second | 7.31 (0.86) | 9.32 (1.80)

23. Secondary Outcome: Pooled Kidney Mass Stage Using 3D CEUS-generated Wash Out Metrics
Description: The association between pooled tumor stage (tumor stages 0,1,2 versus tumor stage 3) and CEUS-generated Wash_Out_Slope parameter was studied. The intensity of the signal (the brightness of the image) is plotted over time to generate the time-intensity curve. The intensity of the signal (the brightness of the image) values range between 0=black, and 255=White. The Wash_Out_Slope decreases as the contrast agent clears the body/mass. Decreasing brightness is related to the slope of the curve. This results in a negative number. This value was generated by fitting the data to a linear equation. Tumor staging is based on the size of the mass, spread to lymph nodes, and metastasis to distant sites according to the AJCC. All masses in this study were in stage 0, I, II, or III (not stage IV). Stage 0 = cancer cell was not found, Stage I = tumor size ≤7 cm, Stage II = tumor size >7 cm, Stage III includes tumors growing into a major vein or tissue, with no spread to lymph nodes.
Time Frame: Baseline- up to 3 minutes
Population: Subjects who complete 3-D CEUS imaging and imaging qualities enough for CEUS parameters calculation.
Measure: Mean (Standard Deviation); unit: AU/second
Groups:
- Non T3: Stage T0, T1 and T2
- Stage T3: Stage T3 disease
Arm/Group | Non T3 | Stage T3
Number analyzed (Participants) | 12 | 2
AU/second | -0.94 (0.16) | -0.87 (0.08)

ADVERSE EVENTS:
Time Frame: 30 minutes post-imaging, up to 1 hour
Groups:
- Perflutren Lipid Microsphere or Lumason: Patients with suspected kidney cancer and planned surgery will be imaged using contrast-enhanced ultrasound. Baseline B-mode US will be performed to confirm the lesions being imaged (unless it is a subject with no lesions, then a basic B-mode US will be performed. 30 minutes post imaging, up to 1 hour.The total imaging time is anticipated to be less than 30 minutes.
Arm/Group | Perflutren Lipid Microsphere or Lumason
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT04021238/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT04021238/ICF_001.pdf